CLINICAL TRIAL: NCT00835016
Title: Early Psychosocial Stimulation (LTP) Program for Children of Depressed Mothers: An RCT
Brief Title: Early Psychosocial Stimulation Program for Children of Depressed Mothers
Acronym: LTP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pakistan Institute of Living and Learning (Other)
Collaborators: The Hincks-Dellcrest Centre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PILL-LTP-0108
Record Dates: First submitted 2009-02-01; First posted 2009-02-03 (Estimated); Last update posted 2020-10-14 (Actual); Status verified 2019-08

CONDITIONS: Maternal Depression; Depression
Keywords: Early psychosocial stimulation, RCT, Depressed mother
MeSH Terms: conditions — Depression | interventions — Long-Term Potentiation; Psychosocial Intervention

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Early psychosocial stimulation (LTP) (Experimental): The 10 session of Early psychosocial stimulation (LTP)will be delivered to depressed mothers in the intervention group
  Interventions: Behavioral: Early psychosocial stimulation (LTP)
- Waiting group (Active Comparator): Waiting group will receive standard follow-up by their own LHWs. This group intervention will be documented at baseline, 3 months (end of the trial) and at 6 months. Similar training of Learning through Play will be provided to the mothers in this group at the end of the study.
  Interventions: Behavioral: Early psychosocial stimulation (LTP)

INTERVENTIONS:
Behavioral: Early psychosocial stimulation (LTP) — Learning through Play (LTP) groups will be conducted weekly for the first eight sessions and two fortnightly sessions. Parenting issues will be discussed with the mothers and play activities will be demonstrated with the children using LTP and home made materials.
  Other Names: Learning Through Play; Psychosocial Intervention for Maternal depression; Randomized Control Trial

SUMMARY:
Aim:

To assess the feasibility of provision of an early psychosocial stimulation programme for the children of depressed mothers and to determine its effect on, mothers depression , mothers' knowledge and practices of childrearing and on children's development.

Hypothesis:

Primary hypothesis:

Mothers attending the psychosocial stimulation program will have significant improvement in the level of depression as compared to the mothers who are on the waiting list.

Secondary hypothesis:

Children of mothers having the intervention will have significantly better growth than the children of mothers who do not have the intervention.

Design:

Randomised controlled trial.

Setting:

An urban slum in a township in Karachi.

Participants:

A total of 130 randomly selected depressed mothers in the intervention group and a total of 130 mothers in the waiting list control group.

Interventions:

Weekly LTP groups for the first eight sessions and two fortnightly sessions. Parenting issues will be discussed with the mothers and play activities will be demonstrated with the children using LTP and homemade materials.

Main outcome measures:

Mothers scores on EPDS & HAM D , Parenting stress as measured by PSI-SF and mothers' knowledge and practices of child rearing measured by questionnaires. Children's height, weight, head and arm circumference.

DETAILED DESCRIPTION:
Research findings suggest that maternal depression affects infant development and growth through multiple processes. Disability due to depressive symptoms (such as fatigue, poor concentration, loss of interest) is likely to affect child-care abilities directly, while impaired social functioning is likely to have indirect consequences through lack of support in childcare. Disturbances in mother-infant relationship in depressed mothers (Cooper 1999) negatively influence the infant's development. The Community-Based Multimodal Psychosocial Intervention LTP has been designed to target these processes and include a supportive component, an educational component (nutritional and healthcare advice)and a parenting programme (Childs psychosocial development through mother-infant play providing stimulation, and support for exploration and autonomy for the infant (Rahman et 2008). The objective will be to help mothers feel supported, empowered and confident about their parenting abilities, and through this process positively influence their mood. Rather than the directive approach of the medical model, health workers will be trained to adopt a more patient-centered approach, tailoring the components according to individual needs of the patient.

Further qualitative testing of the intervention will take place, This will help us to further refine the intervention package, and understand the underlying mediators (maternal mood state, levels of social support, appropriate care, etc) and moderators (education, socioeconomic status) of intervention. Some or all of these important mediators/moderators will then be later studied in detail. Detailed documentation, protocol and training-programme development for the intervention will take place in this trial.

We plan to have this intervention delivered over a three months period. Initially we will deliver weekly sessions in the first 8 weeks of recruitment. This will be followed by two fortnightly sessions in the third month. Thus making a total of 10 sessions. Each session would take up to one hour. These group sessions will be carried out at the health centre.

The trial will give an opportunity to test if the proposed intensity and duration of the intervention are acceptable to participants and to set into place mechanisms to ensure a high level of consistency with which the intervention is delivered. Feedback of performance will give an idea of how frequently refresher training is to be provided and the intervention delivery monitored. Outcome measures for the main trial and cost-effectiveness will also be tested during this phase.

The proposed pilot trial design is a single-blind study, with two parallel groups randomised individually.

ELIGIBILITY:
Inclusion Criteria:

• All Mothers of children aged between 6-30 months having maternal depression

Exclusion Criteria:

* Subjects will not be included in the trial if they have a diagnosed medical condition or significant physical or learning disability, postpartum or other form of psychosis, or are currently under psychiatric care.
* Mothers of children with any serious medical or psychiatric illness will also be excluded.
* The age range of mothers for inclusion in the study will be 16 to 40 years, and all subjects should intend to stay in the study area for at least another 6 months.

Ages: 16 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 260 (Actual)
Dates: Start 2009-02 (Actual); Primary Completion 2010-07 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
The primary outcome measure will be mother's depression scores on EPDS. | change in scores from baseline to 3-month and 6month
  The EPDS is a 10-item symptoms scale for postnatal depression that has been validated in the Pakistani population. Higher scores indicate higher level of depression

SECONDARY OUTCOMES:
Children's height | change in scores from baseline to 3-month and 6-month
  Height measured in cm
Children's weight | Change in scores from baseline to 3-month and 6-month
  Weight measured in kgs
Children's head circumference | Change in scores from baseline to 3-month and 6-month
  Measured in cm
Children's arm circumference | Change in scores from baseline to 3-month and 6-month
  measured in cm
mother's depression score on Hamilton Rating Scale for Depression HAMD | Change in scores from baseline to 3-month and 6-month
  HAMD was used to assess severity of depression, Higher score indicates higher level of dpression.
Mother's scores on Parenting stress Index | Change in scores from Baseline to 3-month and 6-month
  used to assess maternal stress in their role as a parent. Higher scores indicate higher level of stress.
mothers' scores on knowledge, attitude and and practices Questionnaire | Change in scores from baseline to 6-month
  used to assess change in maternal knowledge, attitude and practices. Higher scores indicate higher level of knowledge about child development.

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Nusrat Husain, Principal Investigator — Pakistan Institute of Living and Learning
Locations (1):
- Community Setting, Karachi, Sindh, Pakistan

REFERENCES:
- [Derived] Husain N, Zulqernain F, Carter LA, Chaudhry IB, Fatima B, Kiran T, Chaudhry N, Naeem S, Jafri F, Lunat F, Haq SU, Husain M, Roberts C, Naeem F, Rahman A. Treatment of maternal depression in urban slums of Karachi, Pakistan: A randomized controlled trial (RCT) of an integrated maternal psychological and early child development intervention. Asian J Psychiatr. 2017 Oct;29:63-70. doi: 10.1016/j.ajp.2017.03.010. Epub 2017 Mar 21. PMID 29061430
- See also: This is the link of the organization Pakistan Institute of Learning and Living which is conducting and sponsoring the research — http://pill.org.pk/